CLINICAL TRIAL: NCT01886599
Title: Open-Label, Parallel Group, Multiple-Dose Study to Evaluate the Pharmacokinetics and Safety of Asunaprevir in Subjects With Renal Function Impairment
Brief Title: Study of the Pharmacokinetics and Safety of Asunaprevir in Patients With Kidney Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: AI447-033
Record Dates: First submitted 2013-06-24; First posted 2013-06-26 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2013-11

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — asunaprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Arm A: Subjects with normal renal function (Experimental): Asunaprevir 100 mg tablet by mouth twice daily for 7 days
  Interventions: Drug: Asunaprevir
- Arm B: Subjects with end stage renal disease (Experimental): Asunaprevir 100 mg tablet by mouth twice daily for 7 days
  Interventions: Drug: Asunaprevir
- Arm C: Subjects with mild renal impairment (Experimental): Asunaprevir 100 mg tablet by mouth twice daily for 7 days
  Interventions: Drug: Asunaprevir
- Arm D: Subjects with moderate renal impairment (Experimental): Asunaprevir 100 mg tablet by mouth twice daily for 7 days
  Interventions: Drug: Asunaprevir
- Arm E: Subjects with severe renal impairment (Experimental): Asunaprevir 100 mg tablet by mouth twice daily for 7 days
  Interventions: Drug: Asunaprevir

INTERVENTIONS:
Drug: Asunaprevir
  Other Names: BMS-650032

SUMMARY:
The purpose of the study is to determine how Asunaprevir is handled by the body of subjects with kidney disease compared with subjects with normal kidney function

DETAILED DESCRIPTION:
Primary Purpose:

Other: The purpose of the study is to determine how Asunaprevir is handled by the body of subjects with kidney disease compared with subjects with normal kidney function

ELIGIBILITY:
Inclusion Criteria:

* Group A: Subjects with normal renal function
* Group B: Patients with end stage renal disease
* Group C: Patients with mild renal impairment
* Group D: Patients with moderate renal impairment
* Group E: Patients with severe renal impairment

Exclusion Criteria:

* History of uncontrolled or unstable cardiovascular, respiratory, hepatic, gastrointestinal, endocrine, hematopoietic, psychiatric and/or neurological disease
* Hepatitis B or C
* Human Immunodeficiency Virus (HIV)
* Recent gastrointestinal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-11; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
AUC(TAU) of Asunaprevir assessed using plasma concentrations on Day 7 | 11 time points on Day 7
  Area under the concentration-time curve in one dosing interval [AUC(TAU)] will be calculated from the blood drug concentration versus time curve

SECONDARY OUTCOMES:
Plasma protein binding (PB) of Asunaprevir will be determined from the 1 hour and 3 hour time points post-dose | 1 and 3 hours of Day 7
Maximum observed plasma concentration (Cmax) of Asunaprevir | 30 time points up to Day 10 (blood) and 3 time points up to Day 7 (urine)
  Pharmacokinetic (PK) parameters will be derived from plasma concentration versus time and urinary excretion data (not applicable for subjects who are anuric)
Unbound Maximum observed plasma concentrations (Cmaxu) of Asunaprevir | 30 time points up to Day 10 (blood) and 3 time points up to Day 7 (urine)
  PK parameters will be derived from plasma concentration versus time and urinary excretion data (not applicable for subjects who are anuric)
Time of maximum observed plasma concentration (Tmax) of Asunaprevir | 30 time points up to Day 10 (blood) and 3 time points up to Day 7 (urine)
  PK parameters will be derived from plasma concentration versus time and urinary excretion data (not applicable for subjects who are anuric)
Minimum observed plasma concentration at one dose interval (C12) of Asunaprevir | 30 time points up to Day 10 (blood) and 3 time points up to Day 7 (urine)
  PK parameters will be derived from plasma concentration versus time and urinary excretion data (not applicable for subjects who are anuric)
Minimum observed plasma concentration at Pre-AM dose (Ctrough) of Asunaprevir | 3 time points up to Day 7 (blood) and 2 time points on Days 1 and 7 (urine)
  PK parameters will be derived from plasma concentration versus time and urinary excretion data (not applicable for subjects who are anuric)
Unbound area under the concentration-time curve in one dosing interval [AUC(TAU)u] of Asunaprevir | 30 time points up to Day 10 (blood) and 3 time points up to Day 7 (urine)
  PK parameters will be derived from plasma concentration versus time and urinary excretion data (not applicable for subjects who are anuric)
Area under the concentration-time curve till time of last sampling [AUC(0-T)] of Asunaprevir | 11 (blood) and 2 (urine) time points on Day 7
  PK parameters will be derived from plasma concentration versus time and urinary excretion data (not applicable for subjects who are anuric)
Terminal elimination half life (T-Half) of Asunaprevir | 30 time points up to Day 10 (blood) and 3 time points up to Day 7 (urine)
  PK parameters will be derived from plasma concentration versus time and urinary excretion data (not applicable for subjects who are anuric)
Percent urinary recovery (%UR) of Asunaprevir | 3 time points up to Day 7 (urine)
  PK parameters will be derived from plasma concentration versus time and urinary excretion data (not applicable for subjects who are anuric)
Apparent total body clearance (CLT/F) of Asunaprevir | 30 time points up to Day 10 (blood) and 3 time points up to Day 7 (urine)
  PK parameters will be derived from plasma concentration versus time and urinary excretion data (not applicable for subjects who are anuric)
Unbound apparent clearance (CLU/F) of Asunaprevir | 30 time points up to Day 10 (blood) and 3 time points up to Day 7 (urine)
  PK parameters will be derived from plasma concentration versus time and urinary excretion data (not applicable for subjects who are anuric)
Renal clearance (CLR) of Asunaprevir | 30 time points up to Day 10 (blood) and 3 time points up to Day 7 (urine)
  PK parameters will be derived from plasma concentration versus time and urinary excretion data (not applicable for subjects who are anuric)
Apparent volume of distribution (Vd/F) of Asunaprevir | 30 time points up to Day 10 (blood) and 3 time points up to Day 7 (urine)
  PK parameters will be derived from plasma concentration versus time and urinary excretion data (not applicable for subjects who are anuric)
Accumulation index (AI): Ratio of AUC(TAU) on Day 7 to AUC(TAU) on Day 1 | 22 (blood) and 3 (urine) time points on Days 1 and 7
  PK parameters will be derived from plasma concentration versus time and urinary excretion data (not applicable for subjects who are anuric)
Safety and tolerability endpoints include all AEs and serious AEs, clinical laboratory tests, ECGs, vital signs and physical examination results | Up to Day 15 and until 30 days post discontinuation of dosing
  All recorded adverse events (AEs) will be listed and tabulated by system organ class, preferred term and renal function group. Vital signs and clinical laboratory test results will be listed and summarized by renal function group and time. Any significant physical examination findings and clinical laboratory results will be listed. Electrocardiogram (ECG) readings will be evaluated by the investigator and abnormalities, if present, will be listed

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- United States (3):
  - Orlando Clinical Research Center, Orlando, Florida
  - Davita Clinical Research, Minneapolis, Minnesota
  - New Orleans Center For Clinical Research, Knoxville, Tennessee